CLINICAL TRIAL: NCT02427906
Title: Effect of Transjugular Intrahepatic Portosystemic Shunt on Gut Microbiota and Associated Inflammatory Factors in Cirrhotic Patients
Brief Title: Effect of Transjugular Intrahepatic Portosystemic Shunt on Gut Microbiota in Cirrhotic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Wang Zhu, MD, Medical Doctor, West China Hospital
Other Study IDs: 2014-151; WCH-2014-151 (Other: West China Hospital)
Record Dates: First submitted 2015-04-06; First posted 2015-04-28 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Cirrhosis; Acquired Portal-systemic Shunt Due to Cirrhosis; Hepatic Encephalopathy
Keywords: cirrhosis; gut microbiota; transjugular portosystemic shunt; hepatic encephalopathy
MeSH Terms: conditions — Fibrosis; Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — whole blood, serum，stool
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- TIPS group: patients who have transjugular intrahepatic portosystemic shunt
- Non-TIPS group: patients who have endoscopic variceal ligation

SUMMARY:
The purpose of this study is to determine the effect of transjugular intrahepatic portosystemic shunt on gut microbiota and associated inflammatory factors in cirrhotic patients.

DETAILED DESCRIPTION:
Cirrhosis is associated with qualitative and quantitative changes in the gut microbiota that can potentiate disease progression and complications such as hepatic encephalopathy (HE) and infections. Dysbiosis or altered gut microbiota, due to decreased autochthonous or commensal taxa, has been found in stool and colonic mucosa in cirrhotic patients, which is in turn linked with disease severity and systemic inflammation.

TIPS can decompress the hypertensive portal vein,so that the intestinal congestion can be decrease too. Hence we summarize that TIPS may have effect on gut microbiota and associated inflammatory factors in cirrhotic patients.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients who received TIPS;
* Treatment-naive to TIPS and major operation involving liver such as surgical shunt, hepatic resection and liver transplantation)

Exclusion Criteria:

* Uncontrolled infection or sepsis;
* Hepatobiliary or pancreatic malignancy or biliary obstruction;
* Vital organ dysfunction;
* Administration of antibiotics (after TIPS and 2 weeks before TIPS);
* Cachexia;
* Pregnant or breeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhotic patients undergoing transjugular intrahepatic portosystemic shunt for any indication at West China Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Changes in fecal microbiota | baseline and 6 month

SECONDARY OUTCOMES:
Incidence of hepatic encephalopathy | 6 month
Changes of blood inflammatory parameter including IL-2（interleukin 2）,IL-6,IL-10,IL-8，TNF-α | baseline and 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Wang, PhD, Study Chair — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China